CLINICAL TRIAL: NCT06500637
Title: A Multi-center Double Blind Placebo Controlled Study to Assess the Safety and Efficacy of TB006 for Improving Core Symptoms in Adults With Autism Spectrum Disorder
Brief Title: TB006 for Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rossignol Medical Center (Other)
Collaborators: Autism Discovery and Treatment Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB-RMC
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — TB006

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TB006 (Experimental): TB006 is a humanized immunoglobulin G4 (IgG4) (S228P) type monoclonal antibody that is highly specific and has a high affinity to human Galectin-3 (hGal-3). Galectins are a ubiquitous group of proteins found in a variety of cells, tissues, and extravascular spaces, and are involved in numerous metabolic processes and functions. The galectins preferentially bind to β-galactoside derivatives and can cross-link surface glycoproteins by binding galactose residues. The Gal-3 protein plays an important role in different pathogenic conditions, including neurodegenerative and neuroinflammatory disorders. Serum levels of Gal-3 have been found to be elevated in ASD.
  Interventions: Drug: TB006
- Placebo (Placebo Comparator): Identical IV solution without TB006 product
  Interventions: Drug: TB006

INTERVENTIONS:
Drug: TB006 — TB006 is a humanized immunoglobulin G4 (IgG4) (S228P) type monoclonal antibody that is highly specific and has a high affinity to human Galectin-3 (hGal-3).

SUMMARY:
Multisite 14-week prospective double-blind placebo controlled parallel-group randomized clinical trial with 14-week open-label extension at the end of double-blind treatment phase for placebo subjects. Eligible subjects will be randomized within each site in 2:1 ratio to receive either TB006 or placebo treatment.

DETAILED DESCRIPTION:
A key molecular mechanism implicated in ASD is immune dysregulation and unchecked neuroinflammation marked by increased microglial activation. Galectin-3 (Gal-3), a galactoside-binding lectin, is critical to activation of neuroinflammation resulting in the proliferation of microglia.7 Gal-3 has been shown to be elevated in individuals with ASD. To inhibit Gal-3's contribution to neuroinflammation, Truebinding has developed TB006, a neutralizing monoclonal antibody against Gal-3. Our overall hypothesis is that TB006 will significantly improve core and associated behavioral symptoms of ASD and be well tolerated with no significant adverse effects in adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Autism Spectrum Disorder as defined below by the ADOS or ADI-R.
2. Between 18 and 35 years of age at baseline.
3. English included in the languages in which the individual is being raised.
4. Autism severity of moderate or higher (≥4) under the 7-item clinical global impression-severity scale.
5. Ability to maintain all ongoing complementary, dietary, traditional, and behavioral treatments constant for the study period.
6. Unchanged complementary, dietary, traditional, and behavioral treatments for two months prior to study entry.
7. In males and females of childbearing age, two forms of birth control must be used unless they are not sexually active.
8. A caretaker who will accompany the patient to all procedures and has adequate contact with the participant to complete caregiver questionnaires.

Exclusion Criteria:

1. LGALS3 rs4644 single nucleotide polymorphism with two copies of the Variant-type allele.
2. History of infusion reactions to immunoglobulin product.
3. Significant self-abusive or violent behavior or evidence of suicidal ideation, plan or behavior.
4. Severely affected as defined by CGI-Severity Standard Score = 7 (Extremely Ill).
5. Severe prematurity (<34 weeks gestation) as determined by medical history.
6. Current uncontrolled gastroesophageal disorders.
7. Current or history of liver or kidney disease as determined by medical history and safety labs (See Laboratory Values Monitoring Plan for specific laboratory values).
8. Genetic syndromes.
9. Congenital brain malformations.
10. Active Epilepsy Diagnosis (Epilepsy Diagnosis is defined as History of two or more unprovoked seizures; Patient with a history of epilepsy who have been off medication without seizures for more than two years do not qualify as active epilepsy).
11. Any medical condition that the PI determines could jeopardize the safety of the study subject or compromise the integrity of the data.
12. Significant negative reaction (i.e., fainting, vomiting, etc.) because of a previous blood draw.
13. Failure to thrive or < 5%ile for Body Mass Index or weight at the time of screening.
14. Concurrent treatment with drug that would significantly interact with the investigational product.
15. Allergy or Sensitivity to ingredients in the investigational product or placebo.
16. Evaluation with the NIH Toolbox or BOSCC within 3 months of entering the study.
17. Planned evaluation with the NIH Toolbox or BOSCC during the study.
18. Pregnancy
19. Current DSM-5 diagnosis requiring alternative pharmacotherapy, e.g., Major Depression, Bipolar Disorder, a psychotic disorder (based on clinical assessment assisted by the Child and Adolescent Symptom Inventory).
20. Refusal to comply with the use of birth control if sexually active.
21. Abnormal vital signs (systolic blood pressure > 180 mmHg or < 90 mmHg; heart rate > 120 beats per minute or < 55 beats per minute; temperature > 101.0o F; oxygen saturation < 90%)
22. Prolonged QTc (defined as > 450ms for males and >470ms for female) or any abnormalities felt by the investigator to be of concern.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scores (CARS) | Baseline, Week 8 and Week 14
  The CARS is a measure of autism severity completed by a clinician. Lower Score is Better. Scores range from 15 to 60.

SECONDARY OUTCOMES:
NIH Toolbox | Baseline and Week 14
  The NIH ToolBox is a set of short assessments for neurodevelopmental assessments. Direction of score depends on individual subtest.
Clinical Global Impression Scale (CGI) | Baseline, Week 8 and Week 14
  The CGI measures the overall disease severity and change. It is completed by a clinician. Scores range from 1 to 7. Lower score is better
Social Responsiveness Scale (SRS) | Baseline, Week 8, Week 12 and Week 14
  The SRS is a caregiver report of autism symptoms Lower Score is Better, Scores range from 30 to 90 (T-scores)
Aberrant Behavior Checklist (ABC) | Screening, Weeks 4, 8, 12 and 14
  The ABC is a 58-item consisting five subscales: hyperactivity, irritability, social withdrawal, stereotypic behavior and inappropriate speech in children with developmental disabilities. A higher score indicates more frequent aberrant behaviors.
Major Parental Concerns | Baseline, Week 8, Week 12 and Week 14
  The parent nominates 2 most problematic symptoms. Responses are documented in a standardized format documenting frequency, intensity, and impact of behavior. The overall severity is rated using a CGI type scale.
Ohio State University Clinical Impressions Scale | Baseline and Week 14
  a clinical rating of severity and improvement of 10 autism domains: social interaction, aberrant/abnormal behavior, repetitive/ritualistic behavior, verbal communication, non-verbal communication, hyperactivity/inattention, anxiety/fears, sensory sensitivities, restricted/narrow interests, autism. Severity will be measured at baseline. Each item is rated from 1 (Normal) to 7 (Among the most severe) with a raw score range of 10-70. The raw score will be reported. Higher scores indicate more severe impairment. At the following time points, improvement will be measured. Each item is rated from 1 (Very much improved) to 7 (Very much worse) with a raw score range of 10-70. The raw score will be reported. Higher scores indicate more severe impairment.
Vineland Adaptive Behavior Scale | Baseline, Week 8 and Week 14
  A scale to assess adaptive behavior in children with developmental/intellectual disabilities. This is a 135-item parent-reported measure with ratings in the following domains: communication, daily living skills, and socialization. The frequency of each item is scaled from 0 (Never) to 2 (Usually). For each domain, there are 45 items with a maximum score of 90. Change in each domain will be measured by the change in standard score. Standard scores are calculated from the raw scores and based on age norms. A higher standard score in any domain indicates a higher level of adaptive behavior in that domain. Domain standard scores will be used to get a standard composite score. Change in adaptive behavior will be measured by the change in the standard score. A higher composite score indicates higher overall adaptive behavior ability.

OTHER OUTCOMES:
Galectin-3 levels | Baseline and Week 14
  Gal-3 levels is generally indicative of increased oligomerization and inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, M.D., Ph.D, Study Director — Rossignol Medical Center; Daniel A Rossignol, MD, Principal Investigator — Rossignol Medical Center
Locations (2):
- United States (2):
  - Rossignol Medical Center, Phoenix, Arizona
  - Rossignol Medical Center, Aliso Viejo, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez JI, Kern JK. Evidence of microglial activation in autism and its possible role in brain underconnectivity. Neuron Glia Biol. 2011 May;7(2-4):205-13. doi: 10.1017/S1740925X12000142. Epub 2012 Jul 6. PMID 22874006
- [Background] Garcia-Revilla J, Boza-Serrano A, Espinosa-Oliva AM, Soto MS, Deierborg T, Ruiz R, de Pablos RM, Burguillos MA, Venero JL. Galectin-3, a rising star in modulating microglia activation under conditions of neurodegeneration. Cell Death Dis. 2022 Jul 20;13(7):628. doi: 10.1038/s41419-022-05058-3. PMID 35859075
- [Background] Wang X, Zhang S, Lin F, Chu W, Yue S. Elevated Galectin-3 Levels in the Serum of Patients With Alzheimer's Disease. Am J Alzheimers Dis Other Demen. 2015 Dec;30(8):729-32. doi: 10.1177/1533317513495107. Epub 2013 Jul 2. PMID 23823143
- [Background] Artik A, Kocaman O, Kara H, Tuncer SC. Galectin-3 levels in school aged children with autism spectrum disorder. Int J Dev Disabil. 2022 Dec 1;69(5):757-761. doi: 10.1080/20473869.2022.2150035. eCollection 2023. PMID 37547549